CLINICAL TRIAL: NCT01142583
Title: Canadian Assessment of the Utility of the Treatment Optimization Recommendations in Multiple Sclerosis
Brief Title: A Canadian Study Assessing the Utility of the Treatment Optimization Recommendations in Multiple Sclerosis
Acronym: CanTOR
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: 000107
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple sclerosis; Expanded Disability Status Scale; Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Canadian Multiple Sclerosis Working Group (CMSWG) has developed practical recommendations on how neurologists can assess the status of subjects on disease modifying drugs (DMDs) and decide when it may be necessary to modify treatment in order to optimize outcomes. These recommendations are based on relapses, disease progression as measured by the Expanded Disability Status Scale (EDSS) or EDSS progression, and magnetic resonance imaging (MRI) outcomes. The CMSWG agreed to compare post-treatment relapse rates and severity to baseline rates and severity in each individual subject. The recommended minimum baseline reference time frame needed to assess relapse rate was 2 years prior to treatment initiation. The objective and prospective relapse data should be ideally collected during this reference period. The CMSWG recommended that the following should be taken into consideration when assessing relapse severity: the effect of the relapse on activities of daily living (ADL), the type and number of systems involved (i.e., relapses that are polysymptomatic or that affect the cerebellar/motor systems tend to be more severe), and whether or not a course of corticosteroids was required. The CMSWG also recommended that, prior to considering treatment modification on the basis of progression in disability, progression should be confirmed at 6 months.

The CMSWG's Treatment Optimization Recommendations (TORs) have been retrospectively applied to the 4 year data set from the PRISMS study. Applying the model to subjects after their first year on therapy allowed for accurate prediction of continued disease activity in the form of relapses in the majority of subjects who actually experienced ongoing attacks. The model was less effective in predicting disability progression, but this may well have been due to the low numbers of subjects on treatment progressing over the study period. This observational study used the TOR model to identify subjects as either candidates for therapy optimization or as candidates to maintain current therapy. All subjects were then followed prospectively until re- assessment will be done with this model.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, inflammatory, demyelinating disease of the central nervous system (CNS) and is one of the most common causes of neurological disability in young adults. The neuropathology of the disease is marked by accumulation of leukocytes in the CNS, oligodendrocyte loss, demyelination, axonal atrophy, and neuronal loss. Clinically it is characterized by multi-focal recurrent attacks of neurological symptoms and signs with variable recovery and eventually, the majority of subjects develop a progressive clinical course of MS. The exact cause of MS is unknown, although an autoimmune process has been implicated. Genetic susceptibility plays a role in disease initiation but unidentified environmental factors may also be involved. Three clinical forms of MS are recognized: primary progressive multiple sclerosis (PPMS), secondary progressive multiple sclerosis (SPMS) and RRMS. Primary progressive subjects are characterized by slow and steady accumulation of neurological deficits from onset without superimposed attacks. Subjects with RRMS have exacerbations or relapses with subsequent variable recovery (remission). Secondary progressive multiple sclerosis is characterized by the steady accumulation of significant and persistent neurological deficit with or without superimposed relapses.

In approximately 90% of subjects, the first presentation of MS is an acute, usually reversible episode of CNS dysfunction, referred to as Clinically Isolated Syndrome (CIS). With the advent of MRI, it has become possible to reasonably predict the clinical course of CIS subjects presenting with abnormal MRI findings. The first 5 year follow up study of CIS subjects presenting with abnormal MRI demonstrated a trend for those with more lesions to develop clinically definite MS (CDMS) more frequently, with 92% of those with 4-10 T2 lesions developing CDMS compared to 67% of those with 2-3 T2 lesions. It is also well established that the vast majority of CIS subjects continue to experience ongoing demyelinating disease activity, as evidenced by MRI, even in the absence of a clinical conversion to CDMS.

The introduction of the disease modifying drugs (DMDs) for MS has had a significant impact on the management of those living with this disease. These DMDs are the first agents that have been shown to alter the natural course of relapsing MS. Although there is evidence that the DMDs significantly reduce disease activity, these agents are not "cures" for MS. Thus, many subjects with MS continue to experience disease activity, in spite of treatment with DMDs, including continued relapses, progressive impairment, and ongoing accumulation of MRI disease burden.

OBJECTIVES

Primary objectives:

* To assess if application of the TOR influences clinicians' decisions regarding DMD treatment in the Canadian clinic setting
* To evaluate the perceived utility of the TOR in the DMD treatment decision making process in the Canadian clinic setting

Secondary objective:

* To determine the proportion of subjects meeting a medium or high level of concern according to the TOR in the Canadian Clinic setting.

This was a non-interventional, open-label, observational, multicentric, phase IV study. Subjects were assessed according to the TOR on two occasions over a prospective 12 month observation period. All subjects were assessed according to the TOR at baseline. Subjects were subsequently assessed according to the TOR either at a time-point within the 12-month period when treatment modification is being considered for reasons other than intolerance or at the end of the 12-month observational period. Treatment decisions after each TOR assessment was noted, and perceptions on the utility of the TOR in the decision making process was captured. Additional feedback on the TOR was collected at the end of the observational period through a separate evaluation questionnaire. The assessments that were carried out at baseline and subsequent visits included EDSS history/current status, relapse history/current status, MRI history/current status, cognitive history/current status (if done) and neutralizing antibody (NAb) history/current status (if done).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with duration of RRMS or CIS ≤ 10 yr from onset of symptoms.
* Subjects aged between 18 and 55 years
* Subjects with EDSS score of 0 to ≤ 4.0
* Subjects on consistent therapy with a single DMD (Avonex®, Betaseron®, Copaxone®, Rebif®) for at least 12 months.
* Subjects whose relapse data over the last 12 months was available in the subject's chart
* Subjects whose EDSS data over the last 12 months was available in the subject's chart
* Subjects who were eligible to receive any of the 4 DMDs
* Consecutive subjects were screened until 10 eligible subjects were enrolled (to minimize any selection bias) - Subject was therefore one of 10 consecutive eligible, consenting subjects
* Subjects who had given written informed consent with the understanding that the subject could withdraw consent at any time without prejudice to future medical care

Exclusion Criteria:

* Subject who was not expected to be followed reliably over the next 12 months
* Subjects with concomitant participation in any other studies involving investigational or marketed products
* Subject wo had previously failed DMD therapy and/or switched between therapies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects with either relapsing-remitting multiple sclerosis (RRMS) or a CIS were enrolled from multiple sites across Canada.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2006-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Assessment of history or current status of Expanded Disability Status Score (EDSS) | Baseline to 12 month TOR assessment
Assessment of history or current relapse status | Baseline to 12 month TOR assessment
Assessment of history or current magnetic resonance imaging (MRI) status | Baseline to 12 month TOR assessment
Assessment of history or current cognitive status | Baseline to 12 month TOR assessment
Assessment of history or current status of neutralizing antibodies (NAb) | Baseline to 12 month TOR assessment

SECONDARY OUTCOMES:
Treatment Optimization Recommendation Questionnaire | At the end of the 12 months observational period.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono a division of EMD Canada Inc., an affiliate of Merck KGaA, Darmstadt, Germany